CLINICAL TRIAL: NCT03147846
Title: The Hematologic Impact of Umbilical Cord Milking Versus Deferred Cord Clamping in Premature Neonates. A Randomized Controlled Trial
Brief Title: The Hematologic Impact of Umbilical Cord Milking Versus Deferred Cord Clamping in Premature Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, lecturer, Zagazig University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: milking vs delayed clamping
Record Dates: First submitted 2017-04-29; First posted 2017-05-10 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Delayed Cord Clamping; Umbilical Cord Milking; Preterm Neonates
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: closed envelop method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed cord clamping (Experimental): Keep the baby at the level or below the placenta for 45-60 seconds before clamping the cord.
  Keep the room temperature at 23-25˚C and wrap the baby if possible
  Interventions: Procedure: delayed cord clamping
- cord milking (Active Comparator): Do 4-5 strips from proximal (maternal) end of the cord (as proximal as possible) towards the baby abdomen with thumb and forefinger Wait for 2 seconds between each stripping Keep the baby at the level of placenta
  Interventions: Procedure: cord milking

INTERVENTIONS:
Procedure: delayed cord clamping — delay of cord clamping for 60 seconds
  Arms: delayed cord clamping
Procedure: cord milking — active cord milking 5 times
  Arms: cord milking

SUMMARY:
Comparing the beneficial effect of cord milking versus deferred cord clamping in preterm neonates. A randomized controlled trial

DETAILED DESCRIPTION:
Placental transfusion either by deferred cord clamping or umbilical cord milking became standard care and recommended management especially in preterm deliveries.1 In average, about 80 ml of blood was found to be transferred to the neoborn by one minute after birth.2 This additional blood can afford extra iron and blood volume giving the benefit of less iron deficiency anemia during the first year of life, less need for blood transfusion, less need for vasopressors and less intraventricular hemorrhage (IVH) by 50%.3 Placental transfusion with different techniques proved safety with no significant risks regarding postpartum hemorrhage, polycythemia, jaundice, Apgar score or admission rates.4 Our study aims to compare delayed cord clamping with umbilical cord milking as the best way for placental transfusion for preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

• Gestational age 24 to 34+6 weeks

Exclusion Criteria:

* Category III CTG
* Monochorionic twins
* Significant antepartum hemorrhage
* IUGR or Rh incompatibility

Ages: 24 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
hematological parameters of the premature neonates | 12 months
  first draw and peak hematocrit value and hemoglobin percent, need for inotropes and blood transfusion

SECONDARY OUTCOMES:
composite neonatal morbidities | 12 month
  incidence of intraventricular hemorrhage, necrotizing enterocolitis, retinopathy, jaundice, sepsis , patent ductus arteriosus, etc

CONTACTS AND LOCATIONS:
Overall Officials: Hytham Atia, MD, Principal Investigator — Armed forces hospitals Southern Region KSA
Locations (1):
- Armed Forces Hospital of Southern Region, Khamis Mushait, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atia H, Badawie A, Elsaid O, Kashef M, Alhaddad N, Gomaa M. The hematological impact of umbilical cord milking versus delayed cord clamping in premature neonates: a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Sep 19;22(1):714. doi: 10.1186/s12884-022-05046-7. PMID 36123638